CLINICAL TRIAL: NCT01302717
Title: Impact of Left Ventricular Pacing on Left Ventricular Systolic Function in High-risk Bradycardia Patients
Brief Title: Left Ventricular Pacing to Avoid Cardiac Enlargement Study
Acronym: LVPACE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in enrollment
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Seil Oh, Dr., Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LVPACE
Record Dates: First submitted 2011-02-19; First posted 2011-02-24 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Complete AV Block; Sick Sinus Syndrome
Keywords: Left ventricular pacing
MeSH Terms: conditions — Sick Sinus Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Right ventricular pacing (Active Comparator)
  Interventions: Device: RV pacing
- Left ventricular pacing (Experimental)
  Interventions: Device: LV pacing

INTERVENTIONS:
Device: LV pacing — The left ventricular lead are positioned preferentially at the posterolateral or lateral venous branches of the coronary sinus.
  Arms: Left ventricular pacing
Device: RV pacing — The right ventricular lead are positioned at the right ventricular apex.
  Arms: Right ventricular pacing

SUMMARY:
In this study, the investigators will examine whether left ventricular pacing is superior to right ventricular apical pacing in preventing deterioration of left ventricular systolic function and cardiac remodeling in patients with bradycardia with high risk for development of pacing-induced heart failure.

DETAILED DESCRIPTION:
In this prospective, we will randomly assign 98 patients who need permanent pacemaker due to complete atrioventricular block or sick sinus syndrome to receive left ventricular pacing (49 patients) or right ventricular apical pacing (49 patients). Patients will be paced with temporary pacemaker lead, and only those with paced QRS duration ≥185 ms will be enrolled.

The primary endpoint is left ventricular ejection fraction measured by modified Simpson method at 12 months. The secondary end points include left ventricular systolic end-systolic and diastolic volume, LV strain, NYHA functional class, exercise performance (using treadmill test), quality of life (using SF-36v2), NT-proBNP at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Sinus-node dysfunction or bradycardia due to advanced atrioventricular block
* Paced QRS duration ≥185 ms

Exclusion Criteria:

* Left ventricular ejection fraction < 50 %
* Acute coronary syndrome
* If they had undergone percutaneous coronary intervention or coronary-artery bypass surgery within the previous 3 months
* if they had a life expectancy of less than 1 year
* if they had received a heart transplant

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-04; Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Left ventricular ejection fraction (%) at 12 months | 12 months
  Measured by modified Simpson's method

SECONDARY OUTCOMES:
Left ventricular end-systolic volume (ml) at 12 months | 12 months
  Measured by modified Simpson method
Left ventricular end-diastolic volume (ml) at 12 months | 12 months
  Measured by modified Simpson method
NYHA functional class | 12 months
Functional capacity | 12 months
  measured by treadmill test
NT-proBNP | 12 months
  plasma level

CONTACTS AND LOCATIONS:
Overall Officials: Seil Oh, MD, PhD, Study Chair — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul